CLINICAL TRIAL: NCT02694042
Title: Mission is Remission®: How Can a Disease Self-management Website Change Care?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges and lack of intervention engagement by participants.
Sponsor: IWK Health Centre (Other)
Collaborators: The Hospital for Sick Children (Other); Stollery Children's Hospital (Other); Alberta Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MIR-1018164
Record Dates: First submitted 2015-08-25; First posted 2016-02-29 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Pediatric Crohn's Disease; Pediatric Ulcerative Colitis
Keywords: Pediatric inflammatory bowel disease; Crohn's disease; Ulcerative colitis; Web-based teaching and support; disease self-management; peer support
MeSH Terms: conditions — Pediatric Crohn's disease; Pediatric ulcerative colitis; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mission is Remission® Group (Experimental): Participants in this group will be given access to the Mission is Remission® web-based teaching and support site. They will also be emailed a link to complete online questionnaires at set time points throughout the study.
  Interventions: Behavioral: Mission is Remission®
- Control Group (No Intervention): Participants in this group will continue to receive standard care without access to the Mission is Remission® website. They will also be emailed a link to complete online questionnaires. At the end of the 6 month study period, participants in this group will be given access to the study website.

INTERVENTIONS:
Behavioral: Mission is Remission® — A web-based teaching a support program for adolescents living with inflammatory bowel disease (IBD).
  Arms: Mission is Remission® Group

SUMMARY:
Crohn's disease and ulcerative colitis, known together as inflammatory bowel disease (IBD), are chronic inflammatory conditions of the gastrointestinal tract. Impacts of IBD such as frequent hospital visits, need for surgery and poor growth, can significantly impact a child's social and academic life. Dealing with a chronic disease forces children to rely more heavily on family members for coping strategies to deal with stress. However, a lot of families do not have the resources (emotional or financial) to provide the level of support needed. A self management site called Mission is Remission® has been created to help adolescents and their families deal with the stressors associated with their disease. The site provides a supportive social network that is centred around learning sessions and active forums discussing topics related to disease self-management and coping. This site actively brings together members of the healthcare team and provides support to families who might not be able to travel for additional appointments outside of routine care. The goal of our research is to understand whether the changes this social support will increase disease-specific knowledge, medication adherence, and health-related quality of life. We will also examine whether these changes may reduce some of the demands placed on the Health Care system (e.g., reduced number of calls and visits to gastroenterology (GI) doctors, or time lost from school/work). In addition, this website has been designed to be adapted in the future to other chronic diseases and will help bring healthcare into the digital age.

DETAILED DESCRIPTION:
Background How do health care professionals help children, help themselves? How do patients become active participants in their own care? The prevalence of chronic conditions, such as IBD, is increasing in Canada [1, 2]. Health care systems need to look for sustainable and effective solutions to improve patient care while reducing health care costs. Crohn's disease (CD) and ulcerative colitis (UC), known collectively as IBD, are chronic relapsing and remitting diseases associated with significant medical (i.e., number of hospitalizations, frequent need for surgery, growth failure) and social (i.e., school absences, interference with pursuit of higher education) morbidity [3]. Medical and social morbidity of IBD are intertwined, and take a significant toll on the health-related quality of life (HRQOL) of these patients [4-6].

IBD manifests during childhood or adolescence in 20% to 25% of patients [7]. This is a crucial time in children's development, both physically [8] and emotionally [9]. Children's relationships with family and peers change significantly over the course of their childhood. Normal social development sees children seeking more emotional support from peers over family members in their adolescent years [10]. However, adolescents with IBD do not follow this pattern [11] and tend to seek continued support from family members and rely on parents' coping strategies to deal with stressors [12]. With increased reliance on family support when dealing with a chronic illness like IBD, children may be faced with additional burden when their parents' are not able to offer them the emotional support they need or do not have coping skills that are effective enough to translate into increased care for their children. Despite this, no interventions (to the authors' knowledge) to benefit psychosocial functioning have been specifically studied in pediatric patients or families with IBD.

Current medical intervention tends to focus exclusively on the disease, and does not focus on disease management and coping through self-management skills. Disease self-management involves -the interaction of health behaviours and related processes that patients and families engage in to care for a chronic disease‖ [13]. Studies in both the adult and pediatric chronic illness literature have shown that comprehensive interventions that augment medical treatments with self management therapy, lead to better medical outcomes and better quality of life than care that is strictly medically focused [4-6, 14-24]. These self-management studies are focused on chronic diseases such as diabetes, asthma and rheumatoid arthritis. There have been several small studies of psychological interventions in adult IBD patients with promising results, though issues with design limited the interpretation of the results [25-28]. Disease self-management is more than simple adherence to treatment guidelines - it also incorporates psychological and social management of living with a chronic illness.

-It's something the investigators know intuitively, but it's also supported by evidence: A child's living conditions and experiences - the determinants of health - shape his or her physical health, development, and well-being, affecting not only childhood but the foundation of their health as adults [29, 30].‖ (Stepping it up Report, pg. 23, Health Council of Canada).

Children's experiences (i.e. access to services), can be directly affected through disease self-management. Self-management training is often provided by tertiary care clinics, which includes disease education, and encouragement/support, usually at the time of diagnosis. Most care is given in concentrated sessions during crises times and is in response to a particular problem, which is not the best time to teach self-management skills. Families who are extremely distressed may, in rare cases, receive formal psychological therapy. Although most families receive excellent medical care in the tertiary care centres, the vast majority of patients do not receive comprehensive disease education and self-management therapy. Very few children with IBD receive comprehensive education and self management therapy even when they attend well organized tertiary care clinics.

Geographic and financial concerns often limit access to psychosocial care and information sessions. In most areas of Canada, psychosocial treatment is available through private care. Psychosocial treatment is available for free through public institutions (Canada Health Act, 1984); however, there are long waiting lists and significant time and financial-costs to patients. Parents would have to travel and take time from work, while children would miss school and other related activities, which may further prevent access to treatment. Many families are reluctant to see a psychologist, social worker or psychiatrist due to the social stigma attached to seeking psychotherapy. For some families, the entire process is perceived as blaming them for their problems [31].

In the past 20 years, treatments aimed at teaching parents and children to change their attitudes or behaviour have been developed and evaluated by means of rigorous, randomized trials [32-41]. Although there is strong evidence that these psychosocial treatments work in reducing symptoms and increasing health related quality of life (HRQOL), they are typically delivered only in specialty clinics by highly trained personnel. Few therapists outside of GI clinics will be knowledgeable enough about the disease to effectively help patients and families integrate their psychological and medical care. Evidence from a large meta-analysis has shown that many self-management treatments can be given with as good or better outcomes by paraprofessionals following evidence-based protocols [42]. The use of web-based programs to deliver self-management care has taken off in recent years. Recent meta-analyses have found improved behavioural outcomes for adults using web-based self-management programs [43] and improvements in symptom and disease control for youth with health conditions [44]. Web-based interventions have been found to be comparable to face-to-face treatments [45], and have demonstrated increased social support when programs utilize chat rooms. As Stinson et al. [44] state, many studies have not been able to determine the durability of treatment effects or the cost-effectiveness of these programs. The current research will attempt to address some of these shortcomings.

Based on the lack of access to disease-specific care outside of existing medical intervention, the Mission is Remission® web-based intervention program was created in 2005 as a pilot study, for use by IBD patients and their families. This is a web-enabled evidence based home program of self-management, information, and social support for pediatric IBD patients aged 12-18, with a separate site for their parents. The site was accessed on a restricted-access web site, and participants worked through the program with help of a coach. The coaches worked in collaboration with gastroenterologists, nurses and a psychologist, but the coaches were not medical professionals. This served as an adjunct to routine medical care but not as prescribed medical therapy by the patient's physician or team. This individualized, interactive 12 session program incorporated multi-media tools for disease education and psychological interventions.

The previous research program enrolled two groups of patients-those with inactive disease and those with active disease, and their parents [46]. Remission was induced in patients with active disease before beginning use of the Mission is Remission® site. Although participants demonstrated improvements in main outcome variables such as HRQOL, and Disease Knowledge, there was no true control group in this study such that statements around the effectiveness of the program in comparison to routine or standard care could not be made. Based on lessons learned from the first Mission is Remission® site, a new site was created, which was made possible from an IWK Auxiliary Grant. The expertise of the web-developer, who has been involved in the development of multiple sites for teens, was pivotal in guiding the site's development. The use of social networking, peer support, and parent-to-parent support was optimized through this process.

The proposed research plans to randomize patients to receive either comprehensive care using the Mission is Remission® site or to receive routine care (i.e. regular hospital clinic visits, appointments with clinicians and other specialists as required).

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric IBD patients (approximately 100 patients randomly assigned to the Mission is Remission® group or the wait-list control group) and one of their parents/primary caregivers;
2. Patient is between 12-18 years of age, inclusive;
3. Meets screening criteria for low self-efficacy;
4. Signed informed consent from parent and assent from patient.

Exclusion Criteria:

1. Not English speaking;
2. Children with cognitive impairment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Questionnaire to Assess Self-Efficacy - Changes from baseline | Baseline, 3 months and 6 months
  Adolescents will complete a questionnaire to assess self-efficacy. This will be done at three time points: baseline, 3 months into the study, and at 6 months (at the end of the study).
Questionnaire to Assess Health Related Quality of Life - Changes from baseline | Baseline, 3 months and 6 months
  Adolescents will complete the IMPACT-III questionnaire which is a health-related quality of life questionnaire for pediatric patients with inflammatory bowel disease. The questionnaire will be completed at three time points: baseline, 3 months into the study, and at 6 months (at the end of the study).

SECONDARY OUTCOMES:
Medication Taking Behavior Questionnaire | Baseline, 3 months and 6 months
  Adolescents will complete a"Medication Taking Behavior" questionnaire to look at medication adherence in this patient population.
Questionnaire to Assess Disease Activity | Baseline, 3 months and 6 months
  The Pediatric Crohn's Disease Activity Index (PCDAI) (Hymans, Markowitz, Otley et al., 2005) will be used to assess disease activity in study participants who have Crohn's disease.This measure assesses disease severity, based on subjective items (e.g, patients's report of abdominal pain, stooling pattern, general well-being) and objective data (e.g. weight and height). The Pediatric Ulcerative Colitis Activity Index (PUCAI) (Turner, Otley, Mack et al., 2007) will be completed to assess disease activity in study participants who have ulcerative colitis. This measure also assesses disease severity, based on subjective items (e.g, patients's report of abdominal pain, stooling pattern, general well-being).
Questions to Assess Disease Knowledge | Over the course of 6 months (on average we expect participants in the intervention group to complete a learning module every one to two weeks)
  Experimental group participants will answer 3-6 questions before and after the completion of each learning module in addition to 37 embedded assessment questions. The control group will complete a subset of these questions on two occasions.
Questions to Assess Physical & Social Activity Participation | Baseline, 3 months and 6 months
  Questions from the 2008/2009 National Longitudinal Survey of Children and Youth were modified for use in the current study. This includes questions on participation in school-based activities (sports, clubs, art), as well as participation in activities outside of school. Other questions ask teenagers to report the frequency of computer use, watching television, and playing video games.
Questions to Assess Transition Readiness | Baseline and 6 months
  The Transition Readiness Assessment Questionnaire 5.0 will be administered to determine how ready teenagers are for adult care. Though variance is expected as a function of age, greater gains in transition readiness are expected for intervention group participants.

OTHER OUTCOMES:
Economic Outcome Assessment - Questions to Assess How Having a Child with IBD Affects a Parent's Life | Baseline and 6 months
  Basic questions on the degree to which having a child with IBD affects a parent's life (e.g., work productivity, ability to do regular activities) will be given to parents. This questionnaire contains 5 items, which have been modified from The Work Productivity and Activity Impairment Questionnaire. Other questions have been modified from Coyte and Guerriere (1998)'s Ambulatory Home Care Record, which ask parents about the time taken away from work/home to attend appointments and receive treatment for their child's IBD.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Otley, MD MSc, Principal Investigator — IWK Health Centre

IPD SHARING:
Plan to Share IPD: No
All collected data is self-reported. Participants will be offered the option of receiving a summary of the study results when they are available. These results are presented as group results (not individual).

REFERENCES:
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Bernstein CN, Wajda A, Svenson LW, MacKenzie A, Koehoorn M, Jackson M, Fedorak R, Israel D, Blanchard JF. The epidemiology of inflammatory bowel disease in Canada: a population-based study. Am J Gastroenterol. 2006 Jul;101(7):1559-68. doi: 10.1111/j.1572-0241.2006.00603.x. PMID 16863561
- [Background] Ferguson A, Sedgwick DM, Drummond J. Morbidity of juvenile onset inflammatory bowel disease: effects on education and employment in early adult life. Gut. 1994 May;35(5):665-8. doi: 10.1136/gut.35.5.665. PMID 8200562
- [Background] Devine EC. Meta-analysis of the effects of psychoeducational care in adults with asthma. Res Nurs Health. 1996 Oct;19(5):367-76. doi: 10.1002/(SICI)1098-240X(199610)19:53.0.CO;2-O. PMID 8848621
- [Background] Von Korff M, Gruman J, Schaefer J, Curry SJ, Wagner EH. Collaborative management of chronic illness. Ann Intern Med. 1997 Dec 15;127(12):1097-102. doi: 10.7326/0003-4819-127-12-199712150-00008. PMID 9412313
- [Background] Fall AJ, Henry RL, Hazell T. The use of an interactive computer program for the education of parents of asthmatic children. J Paediatr Child Health. 1998 Apr;34(2):127-30. doi: 10.1046/j.1440-1754.1998.00178.x. PMID 9588633
- [Background] Griffiths AM. Inflammatory Bowel Disease. Adolesc Med. 1995 Oct;6(3):351-368. PMID 10358322
- [Background] Tanner, J., Fetus into Man: Physical growth from conception to maturity, revised edition. 1990, Cambridge, MA: Harvard University Press. 288.
- [Background] Choudhury S, Blakemore SJ, Charman T. Social cognitive development during adolescence. Soc Cogn Affect Neurosci. 2006 Dec;1(3):165-74. doi: 10.1093/scan/nsl024. PMID 18985103
- [Background] Levitt, M.J., N. Guacci-Franco, and J.L. Levitt, Convoys of social support in childhood and early adolescence: Structure and function. Developmental Psychology, 1993. 29(5): p. 811-818.
- [Background] MacPhee M, Hoffenberg EJ, Feranchak A. Quality-of-life factors in adolescent inflammatory bowel disease. Inflamm Bowel Dis. 1998 Feb;4(1):6-11. doi: 10.1097/00054725-199802000-00002. PMID 9552222
- [Background] Gryboski JD. Ulcerative colitis in children 10 years old or younger. J Pediatr Gastroenterol Nutr. 1993 Jul;17(1):24-31. doi: 10.1097/00005176-199307000-00004. PMID 8350209
- [Background] Haynes, R.B., Introduction, in Compliance in Health Care, R. Haynes, D. Taylor, and D. Sackett, Editors. 1979, Johns Hopkins University Press: Baltimore. p. 1-7.
- [Background] Perez MG, Feldman L, Caballero F. Effects of a self-management educational program for the control of childhood asthma. Patient Educ Couns. 1999 Jan;36(1):47-55. doi: 10.1016/s0738-3991(98)00075-5. PMID 10036559
- [Background] Clark NM, Nothwehr F. Self-management of asthma by adult patients. Patient Educ Couns. 1997 Dec;32(1 Suppl):S5-20. doi: 10.1016/s0738-3991(97)00092-x. PMID 9516756
- [Background] Allen RM, Jones MP, Oldenburg B. Randomised trial of an asthma self-management programme for adults. Thorax. 1995 Jul;50(7):731-8. doi: 10.1136/thx.50.7.731. PMID 7570406
- [Background] Holzheimer L, Mohay H, Masters IB. Educating young children about asthma: comparing the effectiveness of a developmentally appropriate asthma education video tape and picture book. Child Care Health Dev. 1998 Jan;24(1):85-99. doi: 10.1046/j.1365-2214.1998.00055.x. PMID 9468782
- [Background] Kolbe J. Asthma education, action plans, psychosocial issues and adherence. Can Respir J. 1999 May-Jun;6(3):273-80. doi: 10.1155/1999/413547. PMID 10393289
- [Background] Bartholomew LK, Czyzewski DI, Parcel GS, Swank PR, Sockrider MM, Mariotto MJ, Schidlow DV, Fink RJ, Seilheimer DK. Self-management of cystic fibrosis: short-term outcomes of the Cystic Fibrosis Family Education Program. Health Educ Behav. 1997 Oct;24(5):652-66. doi: 10.1177/109019819702400511. PMID 9307900
- [Background] Grey M, Boland EA, Davidson M, Yu C, Sullivan-Bolyai S, Tamborlane WV. Short-term effects of coping skills training as adjunct to intensive therapy in adolescents. Diabetes Care. 1998 Jun;21(6):902-8. doi: 10.2337/diacare.21.6.902. PMID 9614605
- [Background] Thoolen B, De Ridder D, Bensing J, Maas C, Griffin S, Gorter K, Rutten G. Effectiveness of a self-management intervention in patients with screen-detected type 2 diabetes. Diabetes Care. 2007 Nov;30(11):2832-7. doi: 10.2337/dc07-0777. Epub 2007 Jul 31. PMID 17666461
- [Background] Ditewig JB, Blok H, Havers J, van Veenendaal H. Effectiveness of self-management interventions on mortality, hospital readmissions, chronic heart failure hospitalization rate and quality of life in patients with chronic heart failure: a systematic review. Patient Educ Couns. 2010 Mar;78(3):297-315. doi: 10.1016/j.pec.2010.01.016. Epub 2010 Mar 3. PMID 20202778
- [Background] Barlow J, Wright C, Sheasby J, Turner A, Hainsworth J. Self-management approaches for people with chronic conditions: a review. Patient Educ Couns. 2002 Oct-Nov;48(2):177-87. doi: 10.1016/s0738-3991(02)00032-0. PMID 12401421
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Schwarz SP, Blanchard EB. Evaluation of a psychological treatment for inflammatory bowel disease. Behav Res Ther. 1991;29(2):167-77. doi: 10.1016/0005-7967(91)90045-5. PMID 2021379
- [Background] Milne B, Joachim G, Niedhardt J. A stress management programme for inflammatory bowel disease patients. J Adv Nurs. 1986 Sep;11(5):561-7. doi: 10.1111/j.1365-2648.1986.tb01288.x. PMID 3534041
- [Background] Garcia-Vega E, Fernandez-Rodriguez C. A stress management programme for Crohn's disease. Behav Res Ther. 2004 Apr;42(4):367-83. doi: 10.1016/S0005-7967(03)00146-3. PMID 14998732
- [Background] Jantschek G, Zeitz M, Pritsch M, Wirsching M, Klor HU, Studt HH, Rasenack J, Deter HC, Riecken EO, Feiereis H, Keller W. Effect of psychotherapy on the course of Crohn's disease. Results of the German prospective multicenter psychotherapy treatment study on Crohn's disease. German Study Group on Psychosocial Intervention in Crohn's Disease. Scand J Gastroenterol. 1998 Dec;33(12):1289-96. doi: 10.1080/00365529850172386. PMID 9930393
- [Background] Sheiham A. Closing the gap in a generation: health equity through action on the social determinants of health. A report of the WHO Commission on Social Determinants of Health (CSDH) 2008. Community Dent Health. 2009 Mar;26(1):2-3. No abstract available. PMID 19385432
- [Background] Raphael D. The health of Canada's children. Part II: Health mechanisms and pathways. Paediatr Child Health. 2010 Feb;15(2):71-6. doi: 10.1093/pch/15.2.71. PMID 21286294
- [Background] Kates N, Craven M, Bishop J, Clinton T, Kraftcheck D, LeClair K, Leverette J, Nash L, Turner T. Shared mental health care in Canada. Can J Psychiatry. 1997 Oct;42(8):suppl 12 pp. doi: 10.1177/070674379704200819. No abstract available. PMID 9417365
- [Background] Saavedra LM, Silverman WK, Morgan-Lopez AA, Kurtines WM. Cognitive behavioral treatment for childhood anxiety disorders: long-term effects on anxiety and secondary disorders in young adulthood. J Child Psychol Psychiatry. 2010 Aug;51(8):924-34. doi: 10.1111/j.1469-7610.2010.02242.x. Epub 2010 Mar 22. PMID 20345838
- [Background] Walco GA, Sterling CM, Conte PM, Engel RG. Empirically supported treatments in pediatric psychology: disease-related pain. J Pediatr Psychol. 1999 Apr;24(2):155-67; discussion 168-71. doi: 10.1093/jpepsy/24.2.155. PMID 10361396
- [Background] Pisterman S, Firestone P, McGrath P, Goodman JT, Webster I, Mallory R, Goffin B. The role of parent training in treatment of preschoolers with ADDH. Am J Orthopsychiatry. 1992 Jul;62(3):397-408. doi: 10.1037/h0079356. PMID 1497105
- [Background] Pisterman S, McGrath P, Firestone P, Goodman JT, Webster I, Mallory R. Outcome of parent-mediated treatment of preschoolers with attention deficit disorder with hyperactivity. J Consult Clin Psychol. 1989 Oct;57(5):628-635. doi: 10.1037/0022-006X.57.5.628. PMID 2794183
- [Background] McGrath PJ, Humphreys P, Keene D, Goodman JT, Lascelles MA, Cunningham JS, Firestone P. The efficacy and efficiency of a self-administered treatment for adolescent migraine. Pain. 1992 Jun;49(3):321-324. doi: 10.1016/0304-3959(92)90238-7. PMID 1408297
- [Background] Feldman W, McGrath P, Hodgson C, Ritter H, Shipman RT. The use of dietary fiber in the management of simple, childhood, idiopathic, recurrent, abdominal pain. Results in a prospective, double-blind, randomized, controlled trial. Am J Dis Child. 1985 Dec;139(12):1216-8. doi: 10.1001/archpedi.1985.02140140050025. PMID 2998181
- [Background] Webster-Stratton C. Advancing videotape parent training: a comparison study. J Consult Clin Psychol. 1994 Jun;62(3):583-93. doi: 10.1037//0022-006x.62.3.583. PMID 8063985
- [Background] Kendall PC. Treating anxiety disorders in children: results of a randomized clinical trial. J Consult Clin Psychol. 1994 Feb;62(1):100-10. doi: 10.1037//0022-006x.62.1.100. PMID 8034812
- [Background] Silverman WK, Kurtines WM, Ginsburg GS, Weems CF, Lumpkin PW, Carmichael DH. Treating anxiety disorders in children with group cognitive-behaviorial therapy: a randomized clinical trial. J Consult Clin Psychol. 1999 Dec;67(6):995-1003. doi: 10.1037//0022-006x.67.6.995. PMID 10596522
- [Background] Manassis K, Mendlowitz SL, Scapillato D, Avery D, Fiksenbaum L, Freire M, Monga S, Owens M. Group and individual cognitive-behavioral therapy for childhood anxiety disorders: a randomized trial. J Am Acad Child Adolesc Psychiatry. 2002 Dec;41(12):1423-30. doi: 10.1097/00004583-200212000-00013. PMID 12447028
- [Background] Weisz JR, Weiss B, Han SS, Granger DA, Morton T. Effects of psychotherapy with children and adolescents revisited: a meta-analysis of treatment outcome studies. Psychol Bull. 1995 May;117(3):450-68. doi: 10.1037/0033-2909.117.3.450. PMID 7777649
- [Background] Wantland DJ, Portillo CJ, Holzemer WL, Slaughter R, McGhee EM. The effectiveness of Web-based vs. non-Web-based interventions: a meta-analysis of behavioral change outcomes. J Med Internet Res. 2004 Nov 10;6(4):e40. doi: 10.2196/jmir.6.4.e40. PMID 15631964
- [Background] Stinson J, Wilson R, Gill N, Yamada J, Holt J. A systematic review of internet-based self-management interventions for youth with health conditions. J Pediatr Psychol. 2009 Jun;34(5):495-510. doi: 10.1093/jpepsy/jsn115. Epub 2008 Nov 23. PMID 19029142
- [Background] Cuijpers P, van Straten A, Andersson G. Internet-administered cognitive behavior therapy for health problems: a systematic review. J Behav Med. 2008 Apr;31(2):169-77. doi: 10.1007/s10865-007-9144-1. PMID 18165893
- [Background] Otley, A.R., P. McGrath, and B. Christensen, The Mission Is Remission(C): a web-enabled self-management program for pediatric IBD targeting health-related quality of life: 158. Journal of Pediatric Gastroenterology and Nutrition, 2005. 41(4): p. 542.
- [Background] Otley, A.R., et al., IMPACT-III is a valid, reliable and responsive measure of health-related quality of life in pediatric Crohn's disease. Journal of Pediatric Gastroenterology and Nutrition, 2006. 43(Suppl 2): p. S49
- [Background] Haaland D, Day AS, Otley A. Development and validation of a pediatric IBD knowledge inventory device: the IBD-KID. J Pediatr Gastroenterol Nutr. 2014 Mar;58(3):313-9. doi: 10.1097/MPG.0000000000000210. PMID 24135980
- [Background] Lipton RB, Stewart WF, Sawyer J, Edmeads JG. Clinical utility of an instrument assessing migraine disability: the Migraine Disability Assessment (MIDAS) questionnaire. Headache. 2001 Oct;41(9):854-61. PMID 11703471
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Hyams JS, Ferry GD, Mandel FS, Gryboski JD, Kibort PM, Kirschner BS, Griffiths AM, Katz AJ, Grand RJ, Boyle JT, et al. Development and validation of a pediatric Crohn's disease activity index. J Pediatr Gastroenterol Nutr. 1991 May;12(4):439-47. PMID 1678008
- [Background] Hyams J, Markowitz J, Otley A, Rosh J, Mack D, Bousvaros A, Kugathasan S, Pfefferkorn M, Tolia V, Evans J, Treem W, Wyllie R, Rothbaum R, del Rosario J, Katz A, Mezoff A, Oliva-Hemker M, Lerer T, Griffiths A; Pediatric Inflammatory Bowel Disease Collaborative Research Group. Evaluation of the pediatric crohn disease activity index: a prospective multicenter experience. J Pediatr Gastroenterol Nutr. 2005 Oct;41(4):416-21. doi: 10.1097/01.mpg.0000183350.46795.42. PMID 16205508
- [Background] Turner D, Otley AR, Mack D, Hyams J, de Bruijne J, Uusoue K, Walters TD, Zachos M, Mamula P, Beaton DE, Steinhart AH, Griffiths AM. Development, validation, and evaluation of a pediatric ulcerative colitis activity index: a prospective multicenter study. Gastroenterology. 2007 Aug;133(2):423-32. doi: 10.1053/j.gastro.2007.05.029. Epub 2007 May 21. PMID 17681163
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Graff LA, Walker JR, Bernstein CN. Depression and anxiety in inflammatory bowel disease: a review of comorbidity and management. Inflamm Bowel Dis. 2009 Jul;15(7):1105-18. doi: 10.1002/ibd.20873. PMID 19161177
- [Background] Statistics Canada. Canadian Internet Use Survey. 2010 [cited 2013 October 28th ]; Available from: http://www.statcan.gc.ca/daily-quotidien/130419/dq130419d-eng.htm.
- [Background] Modi AC, Pai AL, Hommel KA, Hood KK, Cortina S, Hilliard ME, Guilfoyle SM, Gray WN, Drotar D. Pediatric self-management: a framework for research, practice, and policy. Pediatrics. 2012 Feb;129(2):e473-85. doi: 10.1542/peds.2011-1635. Epub 2012 Jan 4. PMID 22218838
- [Background] Bronfenbrenner, U., The Ecology of Human Development: Experiments by Nature and Design. 1979, Cambridge, MA: Harvard University Press.
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391